CLINICAL TRIAL: NCT00334464
Title: A Controlled Clinical Pharmacogenetic Study of a CYP2C9 Plus VKORC1 Polymorphism-Based Individualized Dosing Algorithm for Warfarin to Increase Efficiency of Achieving Therapeutic Dosing
Brief Title: A Pharmacogenetic Study of Warfarin Dosing, "The COUMA-GEN Study"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Deseret Foundation (Other); LDS Hospital Cardiovascular Research (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 128-120
Record Dates: First submitted 2006-06-05; First posted 2006-06-07 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Atrial Fibrillation; Deep Vein Thrombosis; Pulmonary Embolism
Keywords: warfarin metabolism; CYP2C0; anticoagulation; genotyping; DVT; PE
MeSH Terms: conditions — Atrial Fibrillation; Venous Thrombosis; Pulmonary Embolism | interventions — Standard of Care

INTERVENTIONS:
Drug: Standard of care or genotyping dosing of warfarin dosing

SUMMARY:
Anticoagulation with warfarin is a common and potentially hazardous therapeutic intervention. It is a leading cause of iatrogenic bleeding events and, hence, of malpractice claims. There are no good alternatives presently for warfarin anticoagulation, and even when alternatives become available (i.e., ximelagatran), cost, labeling, and experience (outcomes-related) issues will continue to favor an extensive and ongoing use of warfarin. If the present study is able to confirm an advantage for a genotype-driven algorithm, in terms of improved efficiency, therapeutic efficacy, and, especially, safety, then a pharmacogenetics approach to warfarin dosing can be recommended as the basis for an Intermountain Health Care (IHC)-wide quality improvement initiative that should improve patient outcomes, reduce resource use (costs of achieving safe and therapeutic anticoagulation), and reduce adverse clinical events. COUMA-GEN is a prospective, randomized study of patients who are to begin chronic warfarin therapy for specific, qualifying clinical reasons (i.e., atrial fibrillation (AF), deep vein thrombosis (DVT), or post-orthopedic surgery prophylaxis). Qualifying patients will be consented and randomized to an individualized, genotype-based warfarin-dosing regimen or to standard care (without knowledge of genotype). In each study arm, a predicted maintenance dose will be determined. All patients will receive a baseline International Normalized Ratio (INR). For patients in all 3 entry strata, a starting dose of warfarin that is twice the assigned daily maintenance dose (according to the specific treatment arm) will be prescribed on the first and second days, and then the dose will revert to the assigned maintenance dose.

DETAILED DESCRIPTION:
The objectives of this study are to determine

1. whether the pharmacogenetic guided arm can maintain patients a greater time in therapeutic range (TTR - percentage of values in the targeted therapeutic range once a therapeutic INR has been established) without clinical adverse events (i.e., bleeding complications or thromboembolic events),
2. whether the pharmacogenetic guided arm can achieve a higher percentage of therapeutic warfarin levels by days 5 and 8 of therapy (without intervening non-study dose adjustment), and
3. whether the pharmacogenetic guided arm can reduce the need for unplanned dose adjustments and additional INR measurements because of excessive (or insufficient) INR level and clinical adverse events, i.e., bleeding complications or thromboembolic events.

The goal is to achieve >75% TTR in the PG-algorithm arm. Compare proportion of patients reaching therapeutic INR on days 5 and 8 and the subsequent and overall proportion ("time") of INR measurements in therapeutic range (TTR) over 3 months between standard and PG-based arms.

This study will enroll 200 qualifying, consenting patients of either gender, 18 years and above, any ethnicity, with life expectancies > 1 year, beginning on chronic outpatient warfarin therapy for AF, or emergency department/outpatient therapy for spontaneous DVT, or inpatient therapy (and continued for 1 mo) after orthopedic surgery for DVT prevention, or heart failure patients (EF<25% or apical akinesis or left ventricular aneurysm or extensive wall motion abnormality) being started on therapy to reduce the risk of thromboembolism.

ELIGIBILITY:
Inclusion Criteria:

* The patient (male or non-pregnant/non lactating female1) must be > 18 years of age.
* The patient or legally authorized representative must sign a written informed consent, prior to the procedure.
* The potentially eligible patient is at high (post-orthopedic surgery) risk of DVT and the treatment plan will include anticoagulation using warfarin with standard of care follow up including INR assessment.
* The potentially eligible patient is diagnosed with DVT or at high (post-orthopedic surgery) risk of DVT and the treatment plan will include anticoagulation using warfarin with standard of care follow up including INR assessment.
* Patient is diagnosed with atrial fibrillation (AF) and the treatment plan will include anticoagulation using warfarin with standard of care follow up including INR assessment.
* Heart failure patients (EF<25% or apical akinesis or left ventricular aneurysm or extensive wall motion abnormality) in sinus rhythm being started on warfarin to reduce the risk of thromboembolism.
* Women of childbearing potential must be using adequate measures of contraception (as determined by the Investigator) to avoid pregnancy and should be highly unlikely to conceive during the study period.
* Women of childbearing potential must have a negative pregnancy test at screen.

Exclusion Criteria:

* Pregnant and/or lactating women and women of child bearing potential not using acceptable means of contraception.
* Participation in any other clinical trials involving investigational or marketed products within 30 days prior to entry in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-02; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
A comparison of the per-patient percentage of out-of-range INRs (<2, >3) over the observation period of up to 3 months as compared with standard (empiric) dosing of warfarin.

SECONDARY OUTCOMES:
The percentage of out-of-range INRs among patients with at least 1 variant allele
The time within the therapeutic INR range of 2-3 (TTR) over the length of study follow-up
The proportion of patients reaching therapeutic INR on days 5 and 8
The time to first therapeutic INR value
The total number of INR measurements made (for safety, efficiency or dose determination reasons)
The number of adverse clinical events in each group, defined as an INR>3.9, clinical bleeding events more than minor (e.g., bruising), major bleeding events, thromboembolic events, stroke (all-cause), MI, and death (all-cause).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Anderson, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- LDS Hospital, Salt Lake City, Utah, United States